CLINICAL TRIAL: NCT05278507
Title: A Prospective, Randomized Study Comparing Device Performance Characteristics and Safety of Arrow Peripherally Inserted Central Catheters With Arrowga+rd Blue Advanced Protection to Standard Unprotected PICCs
Brief Title: Comparing Arrow PICC Catheters w/ Arrowga+rd Blue Advanced Protection Performance and Safety to Unprotected PICC's
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Teleflex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-10
Record Dates: First submitted 2022-02-21; First posted 2022-03-14 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2022-03

CONDITIONS: Peripherally Inserted Central Catheter
Keywords: PICC

STUDY DESIGN:
Intervention Model Description: The primary purpose of this study is to prospectively collect outcome data in order to evaluate the performance and safety of the Arrowga+rd Blue Advanced PICC with regard to first attempt insertion success and incidence of complications as compared to use of standard, unprotected PICC devices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arrow PICC With Arrowga+rd Blue Advanced Protection (Experimental): The Arrow PICC with Arrowga+rd Blue Advanced protection (Teleflex Medical Incorporated, Morrisville, NC, USA; hereafter referred to as "AGBA") is an FDA-cleared pressure injectable device that offers both antimicrobial and anti-thrombogenic protection for at least 30 days. The application of Arrowga+rd Blue Advanced protection uses a proprietary process whereby chlorhexidine is chemically bonded to the intra- luminal catheter surfaces from tip to hub, and extra-luminal catheter body. The device is cleared for marketing in the United States of America by the Food and Drug Administration, and has obtained the CE mark for marketing in the European Union. The French size and length selected for use will be documented.
  Interventions: Device: Arrowga+rd Blue Advance Protection PICC Placement
- Standard of Care PICC (Sham Comparator): The standard, unprotected PICC currently in use at the institution will be used in this study (here after referred to as Standard). The details of the PICC selected will be recorded including brand, French size, and length.
  Interventions: Device: Sham Comparator PICC placement

INTERVENTIONS:
Device: Arrowga+rd Blue Advance Protection PICC Placement — The PICC will be placed by a qualified healthcare professional, in accordance with institutional policies and procedures and the device's IFU.
  Arms: Arrow PICC With Arrowga+rd Blue Advanced Protection
Device: Sham Comparator PICC placement — The sham comparator PICC will be placed by a qualified healthcare professional, in accordance with institutional policies and procedures and the device's IFU.
  Arms: Standard of Care PICC

SUMMARY:
This study seeks to compare the standard unprotected PICC with the AGBA PICC for placement success, incidence of venous thrombosis through duplex ultrasound, observing for signs and symptoms of thrombotic occlusion and recording treatment response when diagnosed by sluggish fluid flow, inability to aspirate blood and or difficulty/inability to infuse via a lumen or lumens of the catheter. The incidence of catheter-related bloodstream infection will also be tracked during the study.

DETAILED DESCRIPTION:
The primary purpose of this study is to prospectively collect outcome data in order to evaluate the performance and safety of the Arrowga+rd Blue Advanced PICC with regard to first attempt insertion success and incidence of complications as compared to use of standard, unprotected PICC devices.

Patients will receive peripherally-inserted central catheters that are indicated for short or long term peripheral access to the central venous system for intravenous therapy, blood sampling, infusion, pressure injection of contrast media and allows for central venous pressure monitoring. Using randomization, patients will be assigned to receive the institution's standard of care uncoated/unprotected PICC or the study device, the Arrow PICC with Arrowga+rd Blue Advanced Protection

Study Device: Arrow PICC With Arrowga+rd Blue Advanced Protection:

The Arrow PICC with Arrowga+rd Blue Advanced protection (Teleflex Medical Incorporated, Morrisville, NC, USA; hereafter referred to as "AGBA") is an FDA-cleared pressure injectable device that offers both antimicrobial and anti-thrombogenic protection for at least 30 days. The application of Arrowga+rd Blue Advanced protection uses a proprietary process whereby chlorhexidine is chemically bonded to the intra- luminal catheter surfaces from tip to hub, and extra-luminal catheter body. The device is cleared for marketing in the United States of America by the Food and Drug Administration, and has obtained the CE mark for marketing in the European Union. The French size and length selected for use will be documented.

Standard of Care: The standard, unprotected PICC currently in use at the institution will be used in this study (here after referred to as Standard). The details of the PICC selected will be recorded including brand, French size, and length.

Study Design: Prospective, randomized, multicenter study

Number of Subjects: 444 subjects will be enrolled in the study and randomized to receive one of the two PICC devices.

Duration of Subject Study Participation:

Maximum of 92 days, which includes a maximum dwell time of 90 days and follow up 1 to 2 days - 9 days post PICC removal. A subject may remain in the study, with the CVC in place, beyond the expected maximum participant duration (90 days dwell, 1 - 2 day posts removal follow up) if the following conditions are met:

* On day 90 dwell, the subject requires continued PICC access, the assigned PICC remains functional, and it is in the best interest of the subject to continue access via the inserted device.
* It is in the best interest of the subject for the PICC to remain in place, due to health concerns precluding device removal.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ 18 years requiring a PICC
* Patient will remain an inpatient for the entire dwell time
* Ability to comply with study requirements of duplex ultrasound procedures prior to and at the time of PICC removal
* Patients cognitively and physically able to give written consent to participate in the study or patient has a legally authorized representative (LAR) who may give written consent to participate in the study

Exclusion Criteria:

* Current diagnosis of venous thrombosis within the venous tract of the proposed catheter
* Diagnosis of peripheral or central vein stenosis (on proposed insertion side)
* History or diagnosis of veno-occlusive disease
* Diagnosis of superior vena cava syndrome
* Known, pre-existing diagnosis of hypercoagulation disorder unrelated to underlying disease
* Previous enrollment in this study
* Currently pregnant or breast feeding
* Skin condition at or within 15 cm of the proposed catheter insertion site, including signs and symptoms of inflammation, rash, crusts, wounds with drainage, sites of intravenous infusion infiltration or extravasation, hematoma, phlebitis and or thrombophlebitis
* Medical, social, and/or psychological problems precluding subject from study participation
* Known allergy or sensitivity to chlorhexidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Estimated)
Dates: Start 2020-01-16 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
First attempt PICC insertion success | During placement
  rate of first attempt insertion success = number of patients with first attempt insertion /total number of patients *100%
  • First attempt insertion success and number of failed attempts will be documented
PICC Placement Success - Confirmation of tip placement in the lower 1/3 of the superior vena cava at or above the superior vena cava/right atrium junction will be performed by chest x-ray or other tip confirmation system/device and documented. | During placement
  Once the PICC placement is complete, confirmation of catheter tip location in the lower 1/3 of the superior vena cava at or above the superior vena cava/right atrium junction will be performed by chest x-ray or other tip confirmation system/device and documented. Any adjustments to catheter length post-insertion must be performed using sterile technique and maximal barrier precautions. The number of adjustments to the inserted PICC needed to achieve proper tip location will be recorded.
Confirmation of tip patency by aspirating each lumen for brisk blood return and flushing each lumen with at least 10 mL of 0.9% NaCl injection USP | up to 92 days
  Once the PICC placement is complete, the inserter will confirm patency by aspirating each lumen for brisk blood return and flushing each lumen with at least 10 mL of 0.9% NaCl injection USP.
  For inpatients, each lumen will be assessed for patency at least every 12 hours and/or before administration of infusion therapies. Patency assessments will be documented.
  * Patency checks resulting in brisk blood return and ability to flush easily will be considered patent.
  * Patency checks resulting in inability to aspirate blood with ability to flush easily will be documented as a withdrawal occlusion.
  * Patency checks resulting in sluggish flow and/or ability to flush will be documented as a partial occlusion.
  * Patency checks resulting in inability to aspirate blood and inability to flush will be documented as a complete occlusion.
Incidence of catheter related bloodstream infection assessed by laboratory confirmed bloodstream infection | up to 92 days
  Subjects will be assessed for laboratory confirmed bloodstream infection (LCBI) as described below through one day post PICC removal
  LCBI 1 Patient of any age has a recognized pathogen, which is an organism not included on the NHSN common commensal list, identified from one or more blood specimens obtained by a culture or non-culture based microbiologic testing method (excluding organisms identified by testing on sera) AND Organism(s) identified in blood is not related to an infection at another site
  LCBI 2 Patient of any age has at least one of the following signs or symptoms:
  fever (>38.0oC), chills, or hypotension AND Organism(s) identified in blood is not related to an infection at another site AND The same NHSN common commensal is identified by a culture or non-culture based microbiologic testing method, from two or more blood specimens collected on separate occasions.

SECONDARY OUTCOMES:
Incidence of complete loss of catheter function versus the total number of effective catheters placed | up to 92 days
  Incidence of total loss of catheter function = number of total loss of catheter function/number of effective catheter placement
Incidence of catheter-associated external wall thrombosis versus the total number of effective catheters placed | up to 92 days
  Incidence of catheter-related external wall thrombosis = number of patients with catheter-related external wall thrombosis/total number of patients with effective catheter placement
Device performance evaluation | During placement
  Evaluate whether the accessories in the package meet the control requirements of the country and the medical institution, whether the guide wire placement is smooth, whether the catheter placement is smooth, and whether the product is smooth and satisfactory
Evaluation of other safety parameters such as Adverse Events and Device Defects during testing | up to 92 days
  1. Vital signs (temperature (C), heart rate (b.p.m.), respiration rate (b.p.m.) and blood pressure (m.m.Hg) throughout the clinical study period);
  2. Laboratory examination (as appropriate during the evaluation process);
  3. The number and incidence of any related adverse events, severe adverse events during the trial
  4. Number and incidence of any device defects during the test

CONTACTS AND LOCATIONS:
Overall Officials: Xiao H Zhang, Study Chair — Peking University People's Hospital
Locations (5):
- China (5):
  - Beijing Hospital, Beijing, Doncheng District
  - The Fifth Medical Center of Chinese PLA General Hospital, Beijing, Fengtai District
  - Peking University Third Hospital, Beijing, Haidian District
  - The First Medical Center of Chinese PLA General Hospital, Beijing, Haidian District
  - Peking University People's Hospital, Beijing, Xicheng District

IPD SHARING:
Plan to Share IPD: Yes
The Study protocol will be come available after the trademark has been registered to investigators whose proposed research has received IRB/EC approval
Supporting Information: Study Protocol
Time Frame: Permanently after trademark registrations
Access Criteria: Investigators whose proposed research has received IRB/EC approval
URL: https://edc.clinflash.net/